CLINICAL TRIAL: NCT06827340
Title: Multiparametric Whole-Body MRI: a Game Changer in Metastatic Prostate Cancer
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: WB-MRI-2022
Record Dates: First submitted 2025-01-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer (Adenocarcinoma)
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
WB-MRI is a next-generation imaging technique standardized with the first version of MET-RADs-P guidelines.This narrative review aims to analyse the main scientific evidence available in the literature, explaining what WB MRI is and showing its decisive role in metastatic PC.

DETAILED DESCRIPTION:
Prostate cancer ranks among the most prevalent tumours globally. While early detection reduces the likelihood of metastasis, managing advanced cases poses challenges in diagnosis and treatment. Current international guidelines support the concurrent use of 99Tc-Bone Scintigraphy and Contrast-Enhanced Chest and Abdomen CT for the staging of metastatic disease and response assessment. However, emerging evidence underscores the superiority of next-generation imaging techniques including PSMA-PET/CT and whole-body MRI (WB-MRI). This review explores the relevant scientific literature on the role of WB-MRI in metastatic prostate cancer. This multiparametric imaging technique, combining the high anatomical resolution of standard MRI sequences with functional sequences such as diffusion-weighted imaging (DWI) and bone marrow relative fat fraction (rFF%) has proved effective in comprehensive patient assessment, evaluating local disease, most of the nodal involvement, bone metastases and their complications, and detecting the increasing visceral metastases in prostate cancer. It does have the advantage of avoiding the injection of contrast medium/radionuclide administration, spares the patient the exposure to ionizing radiation, and lacks the confounder of FLARE described with nuclear medicine techniques. Up-to-date literature regarding the diagnostic capabilities of WB-MRI, though still limited compared to PSMA-PET/CT, strongly supports its widespread incorporation into standard clinical practice, alongside the latest nuclear medicine techniques.

ELIGIBILITY:
Inclusion Criteria: Literature extracted through the PubMed search engine, following PRISMA checklist, using the keywords:

* "Whole Body MRI"
* "Diffusion Weighted Imaging"
* "PET-CT and WB-MRI"
* "Metastatic Prostate Cancer"
* "Biochemical Recurrence in Metastatic Prostate Cancer"
* "DWIBS"
* "Multiparametric MRI"
* "response assessment in metastatic prostate cancer"
* "Dixon Method",
* "bone biopsy in metastatic prostate cancer",
* "bone metastases in prostate cancer",
* "MET-RADs".
* analysis from 1995 to April 2024.

Exclusion Criteria:

* duplicates
* repetitive,
* irrelevant,
* unrelated,
* out-of-date guidelines,
* case reports

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Literature with patients with metastatic prostate cancer.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 1995-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Identifying the imaging features of metastatic PC in WB-MRI | from 1995 to april 2024
Evaluation of Bone Metastases with WB-MRI | from 1995 to April 2024
Assessment of Nodal Disease | from 1995 to april 2024
Assessment of Visceral Disease | from 1995 to april 2024
Assessing Local Disease and Biochemical Recurrence | from 1995 to april 2024
Response Assessment in Metastatic Prostate Cancer | from 1995 to april 2024

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Bianchi, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No